CLINICAL TRIAL: NCT02359188
Title: Influence of Transcutaneous Vagal Nerve Stimulation on Expression of microRNA, Cytokines, Chemokines and Neuropeptides as Well as Cerebral Resting State and Gastric Motility
Brief Title: Transcutaneous Vagal Nerve Stimulation: Influence on miRNA, Inflammation, Cerebral Resting State and Gastric Motility
Acronym: EpimiRNA_D
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Philipps University Marburg (Other)
Collaborators: European Commission (Other)
Responsible Party: Principal Investigator, Sebastian Bauer, Dr., Philipps University Marburg
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: KKS-207
Record Dates: First submitted 2015-02-04; First posted 2015-02-09 (Estimated); Last update posted 2018-09-13 (Actual); Status verified 2018-09

CONDITIONS: Epilepsy
Keywords: Vagus Nerve Stimulation
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- tVNS (Active Comparator): Transcutaneous vagal nerve stimulation with 25 Hz
  Interventions: Device: Transcutaneous vagal nerve stimulation
- Sham-tVNS (Sham Comparator): Sham transcutaneous vagal nerve stimulation with 1 Hz
  Interventions: Device: Transcutaneous vagal nerve stimulation

INTERVENTIONS:
Device: Transcutaneous vagal nerve stimulation — 4 hours of transcutaneous vagal nerve stimulation
  Other Names: NEMOS tVNS device

SUMMARY:
Randomized, double-blind trial to investigate the influence of a single 4 hours episode of transcutaneous vagal nerve stimulation on the expression of microRNA, various cytokines, chemokines, neuropeptides, cerebral resting state and gastric motility in healthy volunteers.

DETAILED DESCRIPTION:
Transcutaneous vagal nerve stimulation (tVNS) is a non-invasive treatment option for epilepsy. TVNS works via electrical stimulation of the vagal nerve in the outer ear area via two steel electrodes and is performed for about 4 hours per day. Its mechanism of action is unknown. We hypothesize that expression of microRNA (miRNA), and/or release of cytokines, chemokines or neuropeptides is involved in the anticonvulsant activity. TVNS might also influence the cerebral resting state as measured by functional magnetic resonance imaging (fMRI). Due to it's anatomical connections, stimulation of the vagal nerve may furthermore result in altered gastric motility.

This study aims to detect levels of miRNA, cytokines, chemokines and neuropeptides in the blood of healthy volunteers before and after 4 hours of conventional tVNS or sham tVNS. Cerebral resting state and gastric motility will be measured by fMRI.

To this end, 60 healthy volunteers will be recruited and divided into 2 groups. 30 healthy volunteers will be treated with tVNS (25 Hz) for 4 hours (tVNS group). 30 healthy volunteers will be treated with sham tVNS (1 Hz) for 4 hours (control group).

On day 1 of the study, participants will be randomized to one of the two groups. Blood will be drawn from all participants at baseline. Both groups receive a standardized breakfast. TVNS ear electrodes will be put into place for 4 hours without electrical stimulation. Thereafter, blood will be drawn.

On day 2 of the study, blood will be drawn, and all participants receive a standardized breakfast again. Afterwards, tVNS (25 Hz) will be performed in participants of the tVNS group, and sham tVNS (1 Hz) will be performed in participants of the control group. TVNS or sham tVNS end after 4 hours. Blood will be drawn immediately after stimulation end. Thereafter, MRI will be performed in all participants (fMRT resting state, gastric motility). This ends the study for the participant.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years
* Written informed consent

Exclusion Criteria:

* pregnancy
* active implants (like cardiac pacemaker, cochlea implant, implanted VNS)
* contraindications for MRI (e. g. metal fragments, claustrophobia)
* skin lesions in the ara of the left ear conch
* nickel allergy
* drug or alcohol abuse
* current acute disease or medical history of chronic disease
* participant is under legal guardianship

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-08; Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
miRNA expression profile in plasma of healthy persons before and after tVNS as compared to before and after sham tVNS | After 4 hours of VNS

SECONDARY OUTCOMES:
Serum concentrations of different cytokines, chemokines and neuropeptides in healthy persons before and after tVNS as compared to before and after sham tVNS | After 4 hours of VNS
Differences in cerebral microstructural (DTI-MRI) and functional (resting state network, fMR) between tVNS group and control group | After 4 hours of VNS
Differences in gastric motility between tVNS group and control group | After 4 hours of VNS

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian Bauer, Dr., Principal Investigator — Philipps-University Marburg, Dept. of Neurology
Locations (1):
- Philipps-University Marburg, Dept. of Neurology, Epilepsy Center Hesse-Marburg, Marburg, Hesse, Germany